CLINICAL TRIAL: NCT06326814
Title: A First-in-human, Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Ascending Single Doses of SAR443809 in Healthy Adult Subjects
Brief Title: A Study to Test if SAR443809 is Tolerated and Safe When Taken as a Single Dose in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TDU16837; U1111-1298-7281 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SAR443809 and placebo dose 1 Arm (Experimental): 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 1
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 2 Arm (Experimental): 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 2
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 3 Arm (Experimental): 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 3
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 4 Arm (Experimental): 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 4
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 5 Arm (Experimental): 6 participants receiving SAR443809 and 2 receiving placebo, subcutaneous administration dose 5
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 6 Arm (Experimental): Optional: 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 6
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo
- SAR443809 and placebo dose 7 Arm (Experimental): Optional: 6 participants receiving SAR443809 and 2 receiving placebo, intravenous administration dose 7
  Interventions: Drug: Humanized anti-Factor Bb monoclonal antibody; Drug: Placebo

INTERVENTIONS:
Drug: Humanized anti-Factor Bb monoclonal antibody — Pharmaceutical form:Solution for injection-Route of administration:IV and SC routes of administration
  Other Names: SAR443809
Drug: Placebo — Pharmaceutical form:Solution for injection-Route of administration:IV and SC routes of administration

SUMMARY:
Primary objective

* The tolerability and safety of SAR443809 Secondary
* The PK parameters of SAR443809
* The PD activity of SAR443809
* The immunogenicity of SAR443809

DETAILED DESCRIPTION:
Screening: up to 56 days (Day -56 to Day -2). Treatment: 1 day (treatment on Day 1, study observation period from Day -1 to Day 3). Follow-up and end of study: 105 days after IMP administration (follow up visits from Day 5 to Day 78; End of study visit on Day 106). Total study duration for each participant: approximately 23 weeks.

ELIGIBILITY:
Inclusion Criteria: Having given written informed consent prior to undertaking any study-related procedure Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs)/treatment-emergent adverse events (TEAEs) | Baseline up to 23 weeks
Incidence of potentially Clinical laboratory abnormalities | Baseline up to 23 weeks

SECONDARY OUTCOMES:
PK parameters of SAR443809 for IV and SC administrations: Maximum plasma concentration observed (Cmax | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: First time to reach Cmax (tmax | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to tlast (AUClast) | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: Area under the plasma concentration versus time curve extrapolated to infinity (AUC0-∞) | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: Terminal half-life associated with the terminal slope (λz) (t1/2z) | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: Time corresponding to the last concentration above the limit of quantification (Clast tlast) | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: total body clearance of a drug from the plasma calculated by dividing dose by AUC (CL) | Baseline up to 23 weeks
PK parameters of SAR443809 for SC administrations: apparent total body clearance of the SC formulation (CL/F) | Baseline up to 23 weeks
PK parameters of SAR443809 for IV and SC administrations: volume of distribution at steady-state (Vss) | Baseline up to 23 weeks
PK parameters of SAR443809 for SC administrations: apparent volume of distribution at steady-state (Vss/F) | Baseline up to 23 weeks
PK parameters of SAR443809 for SC administrations: absolute bioavailability (F) | Baseline up to 23 weeks
Complement alternative pathway activity (Wieslab AP and alternative pathway hemolytic activity [AH50]) | Baseline up to 23 weeks
  Ex vivo activity of the alternative pathway of complement in serum using the WIESLAB® Complement System Alternative Pathway kit and a hemolytic assay (AH50)
Complement classical pathway activity (Wieslab CP) | Baseline up to 23 weeks
  Ex vivo activity of the alternative pathway of complement in serum using the WIESLAB® Complement System Classical Pathway kit
Incidence of treatment -emergent Anti-SAR443809 antibodies | Baseline up to 23 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Parexel International Site Number : 8400002, Glendale, California
  - Parexel International Site Number : 8400003, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org